CLINICAL TRIAL: NCT06821919
Title: Evaluating the Effect of Hemodialysis Modality and New Anti-glycemic Drugs on NETosis on in Hemodialysis and Diabetic Patient, and Assessment of NETosis in Various Kidney Diseases
Brief Title: Impact of Antiglycemic & Immunosuppressive Therapies on NETosis in Diabetes & Kidney Disease (NETs - Neutrophil Traps)
Acronym: NETs
Status: Recruiting | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Etty Kruzel-Davila, Director of the Nephrology Department, Western Galilee Hospital-Nahariya
Other Study IDs: 0108-22-NHR
Record Dates: First submitted 2025-01-26; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus; Kidney Disease
Keywords: NETosis; Diabetes mellitus; kidney disease; glomerulonephritis
MeSH Terms: conditions — Diabetes Mellitus; Kidney Diseases; Glomerulonephritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples to examine NETosis markers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Diabetes mellitus patients: 2. Diabetic Patients (DM Therapy Study)
  * Sample Size: 20 diabetic patients.
    * Group 1: 10 patients treated with Forxiga/Jardiance (SGLT2 inhibitors).
    * Group 2: 10 patients treated with Ozempic (GLP-1 agonist).
  * Patient Criteria:
    o Patients naïve to SGLT2 inhibitors and GLP-1 receptor agonists to ensure the observed effects are attributable to the initiation of these therapies.
  * Sample Collection:
    * Serum samples (6 ml in serum separator tubes).
    * Two tubes (12 ml total) will be collected per participant at each time point:
  Before starting treatment and at 1, 2, 3, 6, and 12 months after initiating medication.
  * Inclusion Criteria:
    * Diabetic patients aged 18 years or older (men and women).
    * Patients who have not previously received SGLT2 inhibitors or GLP-1 receptor agonists.
  * Exclusion Criteria:
    * Patients with conditions affecting NETosis, including autoimmunity, hematologic or oncologic diseases, or positive for HIV or Hepatitis B/C.
- Chronic kidney disease (CKD) patients: Chronic Kidney Disease (CKD) Patients (Evaluation of Immunosuppressive Therapy)
  * Sample Size: 50 CKD patients with various etiologies.
  * Focus:
    o This part of the study will specifically evaluate immune-mediated kidney disease, such as ANCA-associated vasculitis, and the effects of immunosuppressive therapy on NETosis.
  * Objective:
    * Assess NETosis markers (e.g., cfDNA, Cit-H3, MPO, NE) before initiating immunosuppressive treatment and at 1, 2, 3, 6, and 12 months of therapy.
    * Correlate NETosis dynamics with clinical variables, including disease activity, renal function, and inflammatory markers.
  * Sample Collection:
    o Serum samples (6 ml in serum separator tubes).
    o Two tubes (12 ml total) will be collected per participant at each time point: Before starting treatment and at 1, 2, 3, 6, and 12 months after initiating medication.
  * Exclusion Criteria:
    * Patients with acute infections, hematologic or oncologic diseases, or positive for HIV or Hepatitis B/C.
- 10 healthy participants will be recruited to the control group (for both studies).: Control Group
  * Sample Size: 10 healthy participants.
  * Objective:
    o Serve as controls for both the diabetic and CKD studies.
  * Sample Collection:
  * Two tubes (12 ml total) will be collected per participant
  * Eligibility:
    * Healthy individuals without underlying medical conditions.

SUMMARY:
This study aims to investigate whether new glucose-lowering medications, such as SGLT2 inhibitors (e.g., Forxiga/Jardiance) and GLP-1 receptor agonists (e.g., Ozempic), can reduce NETosis in diabetic patients, thereby mitigating secondary complications such as cardiovascular disease and kidney damage. By targeting dysregulated NET formation, the study seeks to establish a link between reduced NETosis and improved clinical outcomes in diabetes.

Additionally, the study will evaluate the effects of immunosuppressive therapies on NETosis in patients with immune-mediated kidney diseases, such as ANCA-associated vasculitis. By correlating NETosis activity with disease progression and treatment response, this research will assess whether reducing NETosis contributes to better management of inflammation and secondary morbidity in these conditions.

Through these evaluations, the study aims to identify potential therapeutic strategies to improve outcomes in both diabetic and chronic kidney disease populations.

DETAILED DESCRIPTION:
Neutrophil extracellular traps (NETs) are an essential component of the innate immune system, designed to trap and neutralize invading pathogens. NETosis, the process by which neutrophils release decondensed chromatin (DNA and histones) decorated with antimicrobial proteins such as myeloperoxidase (MPO) and neutrophil elastase (NE), is a critical mechanism in host defense. This process is induced by stimuli such as PMA, antibodies, cytokines, chemokines, and sterile triggers, including high glucose, cholesterol, and hypoxia. This stimulation activates the Raf-MEK-ERK pathway and NADPH oxidase-dependent production of reactive oxygen species.1,2 An increase in cytosolic calcium cations activates NADPH oxidases and acts as a cofactor for peptidylarginine deiminase 4 (PAD4). PAD4 catalyzes citrullinated histone H3 (Cit-H3) inducing chromatin decondensation, resulting in a cell extrusion of mixture of DNA and bactericidal proteins, including MPO and NE, which all serves as a specific markers of NETosis.1,2 While beneficial in infection settings, excessive or dysregulated NET formation can cause significant tissue damage and organ dysfunction. NETs have been implicated in the pathogenesis of various acute and chronic inflammatory diseases, including myocardial infarction, atherosclerosis, autoimmune diseases, diabetes, and chronic kidney disease (CKD). Elevated NETosis markers, including cell-free DNA (cfDNA) and Cit-H3, are commonly observed in these conditions, underscoring their role in disease progression.3 Given the dual nature of NETosis, understanding how different factors influence this process is critical for developing targeted therapies. This study focuses on two key aspects: evaluating the effects of antiglycemic medications on NETosis and investigating NETosis across different stages of immune-mediated kidney disease before and after immunosuppressive therapy.

(The hemodialysis part of this trial is not included in the current protocol)

Part 1: Evaluating the Effects of Antiglycemic Medications on NETosis Dysregulated NETosis in diabetic and CKD patients contributes to systemic inflammation and organ damage. Studies have shown elevated levels of NETosis markers, such as cfDNA and Cit-H3, in these populations. While metformin has demonstrated the ability to reduce NET formation in diabetic patients, the effects of newer glucose-lowering agents, including SGLT2 inhibitors and GLP-1 receptor agonists, remain unexplored.4 Both SGLT2 inhibitors and GLP-1 receptor agonists have demonstrated robust cardiovascular and renal protective effects.5 This study aims to evaluate their impact on basal and stimulated NETosis in diabetic and CKD patients with various etiologies. By analyzing NETosis markers before and after treatment, this research will provide insights into whether these agents can modulate NETosis, thereby offering additional anti-inflammatory benefits and reducing disease-associated complications.

Part 2: Evaluating NETosis at Different Stages of Immune-Mediated Kidney Disease and After Immunosuppressive Therapy Immune-mediated kidney diseases, such as ANCA-associated vasculitis, involve heightened NETosis that contributes to kidney injury and systemic inflammation.2 Chronic kidney disease resulting from these conditions often exhibits elevated NET formation, exacerbating disease progression. This study seeks to investigate the dynamics of NETosis at various stages of CKD caused by immune-mediated diseases.

In addition, the effects of immunosuppressive therapy on NETosis will be assessed. Immunosuppressive medications, a cornerstone in the treatment of diseases like ANCA-associated vasculitis, can influence neutrophil activity. By monitoring NETosis markers, including cfDNA, Cit-H3, MPO, and NE, before and after initiating immunosuppressive therapy, the study aims to identify patterns of response and the potential therapeutic modulation of NETosis.

Conclusion This comprehensive investigation into the effects of antiglycemic medications and immunosuppressive therapy on NETosis will provide critical insights into the interplay between treatment, inflammation, and disease progression in diabetic and CKD patients. These findings may help pave the way for targeted interventions aimed at modulating NETosis and improving outcomes in high-risk populations.

ELIGIBILITY:
Inclusion Criteria:

DM therapy study: - Diabetic patients aged 18 years or older (men and women).

* Patients who have not previously received SGLT2 inhibitors or GLP-1 receptor agonists.

  -Chronic kidney disease (CKD) patients :50 CKD patients with various etiologies.

  • Focus:
* This part of the study will specifically evaluate immune-mediated kidney disease, such as ANCA-associated vasculitis, and the effects of immunosuppressive therapy on NETosis.

  • Exclusion Criteria:
* Patients with acute infections, hematologic or oncologic diseases, or positive for HIV or Hepatitis B/C

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: DM therapy study: - Diabetic patients aged 18 years or older (men and women).
  * Patients who have not previously received SGLT2 inhibitors or GLP-1 receptor agonists.
    • Exclusion Criteria:
  * Patients with conditions affecting NETosis, including autoimmunity, hematologic or oncologic diseases, or positive for HIV or Hepatitis B/C.
  Chronic kidney disease (CKD) patients :This study will include 50 CKD patients with various etiologies, with a focus on those with immune-mediated kidney diseases, such as ANCA-associated vasculitis. The primary aim is to evaluate the effects of immunosuppressive therapy on NETosis. All patients will be naïve to prior immunosuppressive therapy to ensure the observed effects are directly attributable to the initiation of treatment.
  • Exclusion Criteria:
  o Patients with acute infections, hematologic or oncologic diseases, or positive for HIV or Hepatitis B/C
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
NETosis marker- citrullinated histone H3 (citH3) | Before treatment, 1,2 , 3, 6 and 12 months after starting anti-diabetic drugs or immunosuppression
  * NETosis markers: NET formation will be assessed in sera blood samples across all groups.
  * Focus on Naïve Patients: Emphasis will be placed on evaluating the initial effects of antiglycemic medications in diabetic patients and the impact of immunosuppressive therapy in CKD patients with immune-mediated diseases.
  * Samples will be collected at identical intervals and compared among diabetic andCKD, groups to assess differences in NETosis levels over time (controls- only baseline NETosis markers) and in response to treatment.
  All serum samples will be diluted 1:2 and citrullinated histone H3 (citH3) will be quantified using the Citrullinated Histone H3 ELISA Kit: O.D. (501620; Cayman Chemical, Ann Arbor, USA).
NETosis marker- Myeloperoxidase | Before treatment, 1,2,3,6 and12 moths after treatment.
  Samples will be collected at identical intervals and compared among diabetic andCKD, groups to assess differences in NETosis levels over time (controls- only baseline NETosis markers) and in response to treatment.
  All serum samples will be diluted 1:2 . MPO measurement will be conducted using Myeloperoxidase ELISA Kit , ng/ml (501410; Cayman Chemical).
NETosis marker- Neutrophil elastase (NE) | Before treatment, 1,2 , 3, 6 and 12 months after starting anti-diabetic drugs or immunosuppression
  Samples will be collected at identical intervals and compared among diabetic andCKD, groups to assess differences in NETosis levels over time (controls- only baseline NETosis markers) and in response to treatment.
  All serum samples will be diluted 1:2 , and NE measurement will be conducted using Human Neutrophil Elastase ELISA Kit, ng/ml (ab204730; Abcam
NETosis marker: Peptidylarginine deiminase 4-PAD4 | Before treatment, 1,2 , 3, 6 and 12 months after starting anti-diabetic drugs or immunosuppression
  Samples will be collected at identical intervals and compared among diabetic andCKD, groups to assess differences in NETosis levels over time (controls- only baseline NETosis markers) and in response to treatment.
  All serum samples will be diluted 1:2 and PAD4 measurement will be conducted using (PADI4 ELISA Kit, ng/ml (ELH-PADI4, RayBiotech) according to the manufacturer's instructions

SECONDARY OUTCOMES:
Kidney function | Before treatment, 1,2 , 3, 6 and 12 months, and each year (during 5 years) after starting anti-diabetic drugs or immunosuppression therapy.
  1. Kidney Function
  * Estimated glomerular filtration rate (eGFR, ml/min) will be measured using CKD-EPI creatinine) equation.
  * These measures will monitor changes in kidney function over time and will be correlated with NETosis markers assessed prior to and during treatment.
Urine protein/ creatinine ratio | Before treatment, 1,2 , 3, 6 and 12 months, and each year (during 5 years) after starting anti-diabetic drugs or immunosuppression therapy
  Urine protein/ creatinine ratio w (mg/gr) will be measured.
  o These measures will monitor changes in kidney function over time and will be correlated with NETosis markers assessed prior to and during treatment
Major adverse cardiovascular events (MACE) | 1,2 , 3, 6 and 12 months, and each year (during 5 years) after starting anti-diabetic drugs or immunosuppression therapy
  Major adverse cardiovascular events (MACE): Including myocardial infarction, stroke, heart failure and cardiovascular death (present/absent).
  * Yearly analyses will evaluate the occurrence of these events in relation to NETosis markers
All cause mortality | 1,2 , 3, 6 and 12 months, and each year (during 5 years) after starting anti-diabetic drugs or immunosuppression therapy
  All-cause mortality: Survival outcomes will be tracked through yearly analyses.
  * Correlations will be drawn between NETosis markers and mortality rates to understand their predictive value and treatment effects. These secondary outcomes will highlight the association between NETosis and long-term renal and cardiovascular outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Galilee Medical Center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Yes
All anonymized data collected during the study will be made available upon reasonable request. This ensures transparency and allows for independent validation of the findings while protecting participant privacy. Identifiable information will be removed, and data will only be shared in a de-identified format, ensuring that participants cannot be traced back based on the shared data. Access to the anonymized dataset will require approval from the principal investigator to ensure appropriate use and adherence to ethical standards.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- Available data/document: Study Protocol: 2022-09-22_012059 — https://my.health.gov.il/CliniTrials/Pages/Home.aspx